CLINICAL TRIAL: NCT00976144
Title: A Single Centre, Randomised, Placebo-controlled, Four-way Cross Over Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK573719 and GW642444 as Monotherapies and Concurrently in Healthy Japanese Subjects
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of GSK573719 (LAMA) and GW642444 (LABA)Administered Individually and Concurrently in Healthy Japanese Subjects
Acronym: DB2113208
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113208
Record Dates: First submitted 2009-09-03; First posted 2009-09-14 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: safety; LAMA; pharmacodynamics; tolerability; Muscarinic receptor antagonist,; anticholinergic,; beta-2 agonist; healthy Japanese subjects; LABA; Chronic Obstructive Pulmonary Disease (COPD); pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK573719, GW642444, GSK573719+GW642444, placebo (Experimental): This is a four-way cross-over study. Subjects, healthy volunteers, will receive a single dose of GSK573719 (500ug), GW642444 (50ug), GSK573719 (500ug)+GW642444 (50ug) administered concurrently, or placebo at each of the four treatment periods. There is a minimum wash-out period of seven days between doses. On enrolment into the study, subjects will be assigned to one of four treatment sequences which are based on a Williams design in accordance with the randomization schedule generated by GSK prior to study start.
  Interventions: Drug: GSK573719

INTERVENTIONS:
Drug: GSK573719 — GSK573719 is a long-acting, inhaled, muscarinic receptor antagonist or anticholinergic bronchodilator. GW642444 is a potent and selective long-acting beta-2 agonist. Both are in development for once daily monotherapies for the treatment of COPD. In this study, their effects are investigated following individual and concurrent administration.
  Other Names: GW642444

SUMMARY:
GW642444 is a potent and selective long-acting beta2 agonist; GSK573719 is a long-acting, inhaled, muscarinic receptor antagonist (or anticholinergic) bronchodilator. Both are in development as once daily (QD) monotherapies for the treatment of Chronic Obstructive Pulmonary Disease (COPD). Development of these two inhaled drugs as a combination therapy is also planned and would have potential for improved efficacy and patient benefit as they both work through different receptor pathways and the combined bronchodilatory effect might be additive.

This study is a randomised, double blind, placebo-controlled, four-way crossover study which will assess the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of GSK573719 and GW642444 in sixteen healthy Japanese subjects. Subjects will receive four possible treatments as single inhaled doses, receiving the two monotherapies separately, the monotherapies concurrently, and placebo.

Blood samples for PK analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of heart rate, blood pressure, ECG and twenty-four hour Holter monitoring, potassium, safety laboratory data and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Japanese ethnic origin defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese.
* Male or female between 20 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until completion of the follow-up visit.
* Body weight > or equal to 45 kg and BMI within the range 18-28 kg/m2 inclusive.
* AST, ALT, alkaline phosphatase and bilirubin < or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block taken from triplicate assessments at screening.
* No clinically active and relevant abnormality on 12-lead ECG or 24h Holter ECG at screening.
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead). A 24hr Holter monitoring recording outside normal limits.
* A history of breathing problems (i.e. history of asthmatic symptomatology, unless asthma in childhood that has now resolved and no longer requires maintenance therapy which should not be an exclusion).
* A mean QTc(B) value at screening >450msec, or an ECG that is not suitable for QT measurements (e.g. LBBB or poorly defined termination of the T wave).
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 40-90 bpm at screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates and benzodiazepines. The detection of drugs with a legitimate medical use would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* A positive test for HIV antibody.
* History of regular alcohol consumption within 3months of the study defined as:

an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). Under Australian guidelines, one standard unit defined as 10g of ethanol, is equivalent to 250ml of full-strength beer, 470 ml of light-strength beer, 100 ml of wine and 30ml of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol. 17. Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products prior to screening.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, tiotropium, atropine and any of its derivatives.
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug.
* The subject has a known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and MgSt.
* Subject is kept under regulatory of judicial order in an institution.
* Any female of childbearing potential.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07-29 (Actual); Primary Completion 2009-09-22 (Actual); Study Completion 2009-09-22 (Actual)

PRIMARY OUTCOMES:
adverse events, cardiac and ECG parameters, vital signs, lung function and clinical laboratory safety assessments | From dosing to 24hr post-dose

SECONDARY OUTCOMES:
plasma concentrations of GSK573719 and GW642444 and derived pharmacokinetic parameters thereof | From dosing to 24 hr post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kelleher DL, Mehta RS, Jean-Francois BM, Preece AF, Blowers J, Crater GD, Thomas P. Safety, tolerability, pharmacodynamics and pharmacokinetics of umeclidinium and vilanterol alone and in combination: a randomized crossover trial. PLoS One. 2012;7(12):e50716. doi: 10.1371/journal.pone.0050716. Epub 2012 Dec 17. PMID 23284643
- See also: Results for study 113208 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113208?search=study&study_ids=113208#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register